CLINICAL TRIAL: NCT00600730
Title: The Effects of Antecedent Hypoglycemia or Exercise on the Response of the Brain to Subsequent Hypoglycemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not available. Could not start this study.
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Steve Davis, Chairman of Medicine, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IRB#040025-Brain and Hypo; R01DK069803-03 (NIH)
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Type 1 Diabetes
Keywords: fMRi; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Hyperinsulinemic euglycemic clamp with fMRi
  Interventions: Procedure: Hyperinsulinemic euglycemic clamp with fMRi
- 2 (Experimental): Hyperinsulinemic hypoglycemic clamp with fMRI
  Interventions: Procedure: Hyperinsulinemic hypoglycemic clamp study with fMRi

INTERVENTIONS:
Procedure: Hyperinsulinemic euglycemic clamp with fMRi — Hyperinsulinemic euglycemic clamp on day 1 with morning fMRi
  Arms: 1
Procedure: Hyperinsulinemic hypoglycemic clamp study with fMRi — Hyperinsulinemic hypoglycemic clamp on day1 with fMRi in morning
  Arms: 2

SUMMARY:
The studies proposed in this application seek to use non-invasive techniques to examine the impact of repeated hypoglycemia on the brain.

DETAILED DESCRIPTION:
The studies proposed in this application seek to use non-invasive techniques to examine the impact of repeated hypoglycemia on the brain.

During the past decade many studies have shown that appropriate magnetic resonance imaging (MRI) methods may be used to assess alterations in brain regional activation in response to external stimuli or tasks. Thus, this non-invasive technique will enhance our ability to learn more about brain function, during hypoglycemia and may delineate information about the role of the brain in hypoglycemia associated autonomic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18-45
* Type 1 diabetes mellitus patients aged 18-45
* Body Mass Index 21-38 kg/m2
* Normal results of routine blood test to screen for hepatic, renal, and hematological abnormalities and an EKG stress test.
* Female volunteers of childbearing potential will undergo HCG pregnancy test. Only women who are not pregnant will participate in the study.

Diabetic Subjects:

* HBA1C= 5.5-11.0%
* Duration of Type 1 Diabetes > 3 yr
* Normal bedside autonomic function

Exclusion Criteria:

All Subjects

* Prior or current history of poor health
* Abnormal results following screening tests
* Pregnancy
* Subjects unable to give voluntary informed consent
* Subjects with a recent medical illness
* Subjects with a history of hypertension, heart disease or cerebrovascular disease
* Subjects with known liver or kidney disease
* Subjects with recent weight loss or consuming a low carbohydrate diet
* Subjects taking steroids
* Subjects taking beta-blockers
* Subjects on anticoagulant drugs, anemic or with known bleeding diatheses
* Evidence of diabetic neuropathy, autonomic neuropathy, proteinuria, extensive background or proliferative retinopathy, hypertension, or cardiovascular disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
fMRi scans | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N Davis, MD, Principal Investigator — Vanderbilt University